CLINICAL TRIAL: NCT04143685
Title: Labor Induction With Misoprostol Versus Oxytocin in Women With Premature Rupture of Membranes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: sammour.rami (Other Government)
Responsible Party: Sponsor-Investigator, sammour.rami, Head of Obstetrics, Bnai Zion Medical Center
Organization: Bnai Zion Medical Center (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MISOX-001
Record Dates: First submitted 2018-12-19; First posted 2019-10-29 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2019-10

CONDITIONS: Prelabor Rupture of Membranes; Premature Rupture of Membrane
Keywords: PROM
MeSH Terms: conditions — Fetal Membranes, Premature Rupture | interventions — Misoprostol; Alprostadil; Oxytocin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- misoprostol (Active Comparator): misoprostol 50 mcg tablet by mouth every four hours for maximum dosage of six
  Interventions: Drug: Misoprostol
- oxytocin (Active Comparator): Oxytocin 10 IU in 1000 mL Standard solution. Starting with 10 mL/hr infusion rate and increasing by 10mL/hr every 20 minutes until achieving 3-5 regular uterine contractions every 10 minutes (as recorded by cardiotocography)
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Misoprostol — Oral administration of cytotec every 4 hours until a maximum of 6 doses
  Other Names: Cytotec; PGE1
  Arms: misoprostol
Drug: Oxytocin — Intravenous infusion of Pitocin through an IVAC until delivery
  Other Names: Pitocin
  Arms: oxytocin

SUMMARY:
This study compares the rate of vaginal delivery after induction of labor with misoprostol versus oxytocin in women with prelabor rupture of membranes. Participants will be randomized to receive either oral misoprotsol every four hours until going into labor, or intravenous oxytocin in increasing dose.

DETAILED DESCRIPTION:
Misoprostol is a synthetic prostaglandin analogue commonly used for labor induction. It causes uterine contractions and ripening of the cervix. Oxytocin sold under the brand name Pitocin among others, is a medication made from the peptide oxytocin and is used to cause contraction of the uterus to start labor.

This randomized controlled trial will compare induction of labor in women with term premature rupture of the membranes and unripe cervix using misoprostol versus oxytocin. The primary outcome is the rate of vaginal delivery. Secondary outcomes will include cesarean section rate, time interval from induction of labor to delivery, neonatal morbidity, patient satisfaction and side effects, as well as chorioamnionitis.

ELIGIBILITY:
Inclusion Criteria:

* Women in their 1st - 4th delivery
* Term prelabor rupture of membranes (37+0 to 42+0 gestational age)
* Vertex presentation
* Singleton pregnancy

Exclusion Criteria:

* Multiple pregnancy
* Previous cesarean section
* Chorioamnionitis on admission
* >2 symptomatic uterine contractions in 10 minutes
* Prostaglandins hypersensitivity
* Contraindication for vaginal delivery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Vaginal delivery rate | During delivery

SECONDARY OUTCOMES:
Operative delivery rate, Cesarean section rate, time interval from induction of labor to delivery | During delivery
chorioamnionitis rate | During or after delivery up to 7 days
  intra-amniotic infection during or after delivery representing in possible combination of maternal fever, fetal tachycardia, maternal leukocytosis, Histopathologic evidence of infection or inflammation or both in the placenta, fetal membranes, or the umbilical cord vessels
Uterine tachysystole | During delivery
Neonatal morbidity | After delivery until discharge
  Apgar score, , ,
Neonatal morbidity | immediately after delivery
  Umbilical Cord Blood Gases
Neonatal morbidity | up to 7 days after delivery
  NICU admission
Neonatal morbidity | up to 7 days after delivery
  Antibiotic administration

CONTACTS AND LOCATIONS:
Locations (1):
- Bnai Zion Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No